CLINICAL TRIAL: NCT04167800
Title: Effects of Exercise Therapy in Addition to Compression Orthotics in Patients With Pectus Carinatum
Brief Title: Effects of Exercise Therapy on Pectus Carinatum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-14/11
Record Dates: First submitted 2019-11-04; First posted 2019-11-19 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Pectus Carinatum
Keywords: Pectus Carinatum; orthosis; exercise
MeSH Terms: conditions — Pectus Carinatum; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): All patients will be instructed to wear the device for 23 weeks for 12 weeks after being instructed on how to use the appropriate compression orthosis. The patient's relatives will be asked to keep a book in order to monitor their use. Patients who have not used the device for 5 consecutive days will be excluded from the study. The first group will be given awareness training on using one session orthosis and posture correction.
- Exercise Group (Active Comparator): In addition to the applications to the first group, mobilization, strengthening, posture and segmental breathing exercises will be given . All of these exercises will be combined with segmental breathing exercises depending on the location of the PC. Exercise therapy will be administered by a physiotherapist with 20 years of experience once a week and will be designed as a home program on the remaining days and will be asked to do 45 minutes twice a day (at least 4 times a week). The patient's relatives will be asked to keep a book to monitor the exercise. Patients who do not perform 5 consecutive exercise sessions will be excluded from the study. All treatments will be given for 12 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Orthosis, mobilization, strengthening, posture and segmental breathing exercises
  Arms: Exercise Group

SUMMARY:
Pectus Carinatum (PC); deformity in which the front wall of the chest protrudes forward. Non-invasive treatment approaches for PC include compression orthosis and exercises that target the deformity itself and concurrent postural impairment and scoliosis. In addition, the formation of muscles can help close the deformity. Although exercise training is recommended, there is no randomized study showing its effectiveness in the literature. Therefore, in our study, the investigators aimed to investigate the effectiveness of exercise therapy in addition to compression orthotics.

DETAILED DESCRIPTION:
A chest wall deformity is a structural abnormality of the chest that can range from mild to severe. Chest wall deformities occur when the cartilage that connects the ribs grows unevenly. It is not clear why this happens, but the condition tends to run in families. The two most common types of chest wall deformity are Pectus excavatum and Pectus carinatum, Pectus carinatum goes far beyond a simple esthetical problem. It can be responsible of physical signs and symptoms and also has significant psychological impact. Defects tend to worsen during pubertal growth spurts and even during adult life. Recent evidence shows that these patients are at risk for a disturbed body image and reduced quality of life and many patients refer feelings of discomfort, shame, shyness, anxiety, anguish, and even depression, which can lead to social isolation. Chest pain or discomfort, especially when lying in prone position, intolerance to physical exercise, scoliosis, impaired shoulders and kyphotic position are some of the physical signs and symptoms.Non-invasive treatment approaches for PC include compression orthosis and exercises that target the deformity itself and concurrent postural impairment and scoliosis. In addition, the formation of muscles can help close the deformity. Most evidence of non-invasive treatment is retrospective or prospective case series. In a prospective case series, patients were instructed to perform chest wall strengthening exercises, but the effects of the exercises were not investigated . Although, exercise training is recommended, there is no randomized study showing its effectiveness in the literature. Therefore, in our study, the investigators aimed to investigate the effectiveness of exercise therapy in addition to compression orthotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PC by doctor and indicated for the first time orthotic use
* A correction pressure of less than 10 pounds per square inch in the compression test
* 10-18 years old,
* Discontented with this deformity

Exclusion Criteria:

* Previous orthosis use
* Severe scoliosis (Cobb angle above 20 degrees)
* Having chronic systemic disease
* Having serious psychiatric illness
* Having complex mixed pectus deformity

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Pectus severity index | Change from Pectus severity index at 12 weeks
  Thorax-caliper measurement: Pectus severity index (T.I.): (T3/T1) * 100 (%), T1: upper edge of the manubrium, T2: Angulus Ludovici, T3: deepest point of the funnel chest, Pectus carinatum: T.I. > 140.
patient's perception of deformity | Change from patient's perception of deformity at 12 weeks
  patient's perception of deformity (0-10): The subject's self-perception of pectus carinatum was obtained through self-report using a scale from 0 (worst self-perception of pectus carinatum) to 10 (best self-perception of pectus carinatum).
Global Rating of Change Score | through study completion, an average of 12 weeks
  The responses for the Global Rating of Change Score is"much better (2)"; "slightly better(1)"; "stayed the same (0)";"slightly worse (-1)" or "much worse (-2)".
Chest anthropometric measurement-1 | Change from baseline the extent of maximal protrusion at 12 weeks
  The extent of maximal protrusion:distance from the point of maximum protrusion to the estimated normal level of chest wall (milimeter).

SECONDARY OUTCOMES:
New York Posture Rating Chart for posture assessment | Change from baseline score of New York Posture Rating Chart at 12 weeks
  The scores of the remaining 10 body alignment segments are summed, allowing a range ofoverall score between 0 and 100, with a score of 100 representing ideal posture
The Nuss Questionnaire modified for Adults (Patient Form) | Change from baseline score of The Nuss Questionnaire modified for Adults (Patient Form) at 12 weeks
  Disease-specific health-related quality of life assessment tool for patients with pectus The patient version of the NQ-mA includes 12 items, scored 1 to 4. Possible minimum and maximum scores are 12 and 48 in the patient form; higher scores indicate a better quality of life.
Chest anthropometric measurement-2 | Change from baseline craniocaudal length at 12 weeks
  Craniocaudal length: craniocaudal length of protruding zone, measured through the point of maximal protrusion
The Nuss Questionnaire modified for Adults (Parent Form) | Change from baseline score of The Nuss Questionnaire modified for Adults (Parent Form) at 12 weeks
  Disease-specific health-related quality of life assessment tool for patients with pectus parent. The parent version of the NQ-mA includes 11 items, scored 1 to 4. Possible minimum and maximum scores are 11 and 44 in the parent form; higher scores indicate a better quality of life.
Chest anthropometric measurement-3 | Change from baseline lateral length at 12 weeks
  Lateral length: length of protruding zone, again measured through the point of maximum protrusion in the transverse direction

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Mehmet Ali Aydınlar University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, ICF will be shared with the authors every two months
Supporting Information: Study Protocol, ICF
Time Frame: Every 2 months
Access Criteria: Must be an author

REFERENCES:
- [Background] Akkas Y, Gulay Peri N, Kocer B, Gulbahar G, Baran Aksakal FN. The prevalence of chest wall deformity in Turkish children. Turk J Med Sci. 2018 Dec 12;48(6):1200-1206. doi: 10.3906/sag-1807-180. PMID 30541247
- [Background] Bahadir AT, Kuru P, Afacan C, Ermerak NO, Bostanci K, Yuksel M. Validity and reliability of the Turkish version of the nuss questionnaire modified for adults. Korean J Thorac Cardiovasc Surg. 2015 Apr;48(2):112-9. doi: 10.5090/kjtcs.2015.48.2.112. Epub 2015 Apr 5. PMID 25883894
- [Background] Banever GT, Konefal SH, Gettens K, Moriarty KP. Nonoperative correction of pectus carinatum with orthotic bracing. J Laparoendosc Adv Surg Tech A. 2006 Apr;16(2):164-7. doi: 10.1089/lap.2006.16.164. PMID 16646710
- [Background] Canavan PK, Cahalin L. Integrated physical therapy intervention for a person with pectus excavatum and bilateral shoulder pain: a single-case study. Arch Phys Med Rehabil. 2008 Nov;89(11):2195-204. doi: 10.1016/j.apmr.2008.04.014. PMID 18996250
- [Background] Ewert F, Syed J, Wagner S, Besendoerfer M, Carbon RT, Schulz-Drost S. Does an external chest wall measurement correlate with a CT-based measurement in patients with chest wall deformities? J Pediatr Surg. 2017 Oct;52(10):1583-1590. doi: 10.1016/j.jpedsurg.2017.04.011. Epub 2017 Apr 27. PMID 28499711
- [Background] Haje SA, Bowen JR. Preliminary results of orthotic treatment of pectus deformities in children and adolescents. J Pediatr Orthop. 1992 Nov-Dec;12(6):795-800. doi: 10.1097/01241398-199211000-00018. PMID 1452753
- [Background] Kravarusic D, Dicken BJ, Dewar R, Harder J, Poncet P, Schneider M, Sigalet DL. The Calgary protocol for bracing of pectus carinatum: a preliminary report. J Pediatr Surg. 2006 May;41(5):923-6. doi: 10.1016/j.jpedsurg.2006.01.058. PMID 16677884
- [Background] Lee RT, Moorman S, Schneider M, Sigalet DL. Bracing is an effective therapy for pectus carinatum: interim results. J Pediatr Surg. 2013 Jan;48(1):184-90. doi: 10.1016/j.jpedsurg.2012.10.037. PMID 23331813
- [Background] Martinez-Ferro M, Bellia Munzon G, Fraire C, Abdenur C, Chinni E, Strappa B, Ardigo L. Non-surgical treatment of pectus carinatum with the FMF(R) Dynamic Compressor System. J Vis Surg. 2016 Mar 17;2:57. doi: 10.21037/jovs.2016.02.20. eCollection 2016. PMID 29078485